CLINICAL TRIAL: NCT06221878
Title: Analysis of the Prognostic Impact of Laparoscopic Surgery in Patients With Systemic Obesity and Colorectal Malignant Tumors
Brief Title: Comparison of Laparoscopic and Open Surgery for Colorectal Malignancy in Obese Patients
Acronym: LOSCRO
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202301534B0
Record Dates: First submitted 2024-01-12; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 1995-01

CONDITIONS: Colorectal Cancer; Obesity
Keywords: Colorectal cancer; obesity; laparoscopy surgery; open surgery; postoperative survival analysis
MeSH Terms: conditions — Colorectal Neoplasms; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic Group: Individuals with a body mass index of ≥ 30 kg/m2 underwent laparoscopic surgery for primary stage I-III colorectal adenocarcinoma.
- Open Group: Individuals with a body mass index of ≥ 30 kg/m2 underwent open surgery for primary stage I-III colorectal adenocarcinoma.

SUMMARY:
The goal of this observational study is to compare laparoscopic and open surgery outcomes in colorectal cancer patients with BMI ≥ 30 kg/m2 . The main question[s] it aims to answer are:

1. the short-term outcome and postoperative outcomes of patients treated with open group versus laparoscopy group
2. the long-term oncologic outcome of patients treated with open group versus laparoscopy group

This study is a retrospective and observational study. Subjects were not be given or offered any treatment during the study. The investigator reviewed the patient's medical history and examination report to determine eligibility based on inclusion and exclusion criteria.

If there is a comparison group: Researchers compared the open group and laparoscopy group to see if the laparoscopic group have better short-term outcomes with comparable oncologic outcomes to the open group.

DETAILED DESCRIPTION:
This study is a retrospective and observational study. Subjects were not be given or offered any treatment during the study. The investigator reviewed the patient's medical history and examination report to determine eligibility based on inclusion and exclusion criteria.

Given the uncertainty regarding the long-term outcomes of laparoscopy in obese patients with CRC, this study aimed to analyse a decade of data comparing laparoscopic and open surgery outcomes in patients with BMI ≥ 30 kg/m2 who had undergone treatment for CRC at the Linkou Chang Gung Hospital.

ELIGIBILITY:
Inclusion Criteria:

* CRC patients with BMI ≥ 30 kg/m2 who underwent colorectal surgery at the Linkou branch of the Chang Gung Memorial Hospital (CGMH) between January 2009 and December 2019.

Exclusion Criteria:

* non-adenocarcinoma neoplasms
* Stage IV CRC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage I ~ III Colorectal adenocarcinoma patients with BMI ≥ 30 kg/m2 who underwent colorectal surgery at the Linkou branch of the Chang Gung Memorial Hospital (CGMH) between January 2009 and December 2019.
Sampling Method: Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Short-term outcome | 2009 to 2019
  Postoperative mortality risk
Short-term outcome | 2009 to 2019
  Postoperative morbidity risk
Short-term outcome | 2009 to 2019
  Clavien-Dindo classification
Short-term outcome | 2009 to 2019
  Length of hospital stay
Short-term outcome | 2009 to 2019
  Incidence of readmission

SECONDARY OUTCOMES:
Long-term Oncologic outcome | 2009 to 2019
  Disease-free survival (DFS)
Long-term Oncologic outcome | 2009 to 2019
  Overall survival (OS)
Long-term Oncologic outcome | 2009 to 2019
  Recurrence rate

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available from the corresponding author upon reasonable request

REFERENCES:
- [Derived] Hsu YJ, Yu YL, Jhuang JR, You JF, Liao CK, Tsai WS, Pan YP, Chern YJ. Comparison of laparoscopic and open surgery for colorectal malignancy in obese patients: a propensity score-weighted cohort study. Int J Surg. 2024 Aug 1;110(8):4598-4607. doi: 10.1097/JS9.0000000000001536. PMID 38833348